CLINICAL TRIAL: NCT02284620
Title: Continuous Femoral Nerve Block Versus Local-wound Infiltration Analgesia For Patients Receiving Unilateral Total Knee Arthroplasty --- A Randomized Controlled Trial
Brief Title: Continuous Femoral Nerve Block Versus Local-wound Infiltration Analgesia For Patients Receiving Total Knee Arthroplasty --- A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, The Department of Anesthesia and Pain Medicine, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYYYMZ-001
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Postoperative Pain; Total Knee Arthroplasty
Keywords: anesthesia; nerve block; infltration
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CFNB group (Experimental): Particiants in this group will receive a single injection for femoral nerve block intra-operatively combined continuous femoral nerve block post-operatively. This technique will be guided by ultrasound and nerve stimulator.The regimen is a loading dose of 0.8% ropivacaine 30 ml intra-operatively and 0.15% ropivacaine 300ml in the form of continuous femoral nerve block post-operatively.
  Interventions: Procedure: CFNB group
- LWI group (Active Comparator): Particiants in this group will receive a peri-articular injection of suspension (48 ml of 0.8% ropivacaine with 2 ml of 40mg methylprednisolone) combined with intravenous patient controlled analgesia post-operatively (tramadol 800 mg and flurbiprofenaxetil 100 mg with saline added up to a volume of 80 ml )
  Interventions: Procedure: LWI group

INTERVENTIONS:
Procedure: CFNB group — CFNB :A single injection of ropivacaine 30ml for femoral nerve block pre-operatively +0.15% ropivacaine 300ml for continuous femoral nerve block post-operatively guided by ultrasound and nerve stimulator.
  Arms: CFNB group
Procedure: LWI group — LWI: 48 ml of 0.8% ropivacaine with 2 ml of 40mg methylprednisolone for intra-articular and peri-articular wound infiltration intra-operatively in combination with intravenous patient controlled analgesia post-operatively.
  Arms: LWI group

SUMMARY:
Post-operative pain after total knee arthroplasty is usually severe and impair the functional recovery of operated joints.The purpose of this study is to determine whether post-operative continuous femoral nerve block analgesia is superior to local wound infiltration combined with intravenous patient controlled analgesia in improving joint function and reducing the incidence of chronic post-surgical pain (CPSP).

DETAILED DESCRIPTION:
Major surgical types for knee included arthroscopy, total or partial knee arthroplastic surgery. These procedures are typically associated with severe pain. Function training, which is imperative after surgery for these patients, also aggravated pain.Post-operative pain after major knee surgery impaired post-operative knee recovery and prolonged inpatient length of stay.To maximize the efficacy and minimize the side effects of different options,a multi-modal analgesic regimen was recommended for patients underwent knee surgeries.Local wound infiltration and nerve block are given considerable attentions.Compared with systematic analgesia,nerve block with local anesthetics has been revealed to provide superior analgesia and better recovery of joint function compared with systemic analgesics. Currently,systematic evidence is sparse related to the comparative efficacy of pain control between local wound infiltration and nerve block,the investigators therefore conduct this randomized controlled trials.

This study was approved by the institutional review board of the First Affiliated Hospital of Chongqing Medical University. The protocol design is in accordance with Consolidated Standards of Reporting Trials (CONSORT) statement . This study is designed as a randomized controlled trial to compare the analgesic efficacy of continuous femoral nerve block (group CFNB) with local wound infiltration (group LWI).

Participants in group CFNB will receive a single injection for femoral nerve block intra-operatively combined with continuous femoral nerve block post-operatively guided by ultrasound and nerve stimulator.

Participants in group LWI will receive a peri-articular injection of suspension (48 ml of 0.8% ropivacaine with 2 ml of 40mg methylprednisolone) combined with intravenous non-opioid patient controlled analgesia.All participants will receive unified post-operative rehabilitation programme and the prophylaxis of infection and thrombo-embolism.

The primary outcome of this study is the incidence of chronic moderate-to-severe post-surgical pain.The secondary outcomes of this study are acute post-operative pain and rescue medication;knee function measured by WOMAC knee scores ;life ability measured by EQ-5D questionnaire;adverse events associated with the post-operative analgesia.

This study will be conducted under the supervision of an independent auditor. Every week, the auditor checked the data of the participants the day after the survey was conducted. Assessment of pain intensity and prognostic outcomes must be confirmed by the auditor in sampled population. When there is disagreement between surgeon and anesthesiologists in evaluating the prognosis of patients, the auditor must solve this disagreement by discussion with both evaluators. Data were double-entered by two statisticians with limitation of access and locked during statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* men and women over the 18 years and younger than 75 years old who had received selective unilateral knee replacement.

Exclusion Criteria:

* bilateral knee replacement
* the secondary knee revision and knee surgery not interfering with articular joint cavity (wound debridement and suture)
* American Society of Anesthesiology (ASA) classification of anesthesia risk IV and V grade; body mass index higher than 35
* coagulation dysfunction, which is assessed by activated partial thromboplastin time (APTT) higher than the upper limit by 10s
* prothrombin time (PT) higher than the upper limit by 5s
* International Normalized Ratio (INR) higher than 1.3, or any of criteria met above
* local infection of puncture sites
* neurological diseases
* uncontrolled general infection
* intra-operative cardiac arrest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
chronic moderate-to-severe post-surgical pain | 3 months post-operatively
  chronic moderate-to-severe post-surgical pain will be measured as more than 3 by numerical rating scale for pain

SECONDARY OUTCOMES:
acute pain post-operatively | Post-operative day 1 to 3
  Pain intensity will be measured by visual analogue scale
Analgesic Rescue | Post-operative day 1 to 3
  The dosages of opioid or non-opioid analgesic rescue medications
Knee function | 3 months ,6 months and 12 months post-operatively
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores will be used.
Life Quality | 3 months ,6 months and 12 months post-operatively
  It will be assessed by EuroQol 5-Dimension Questionnaire(EQ-5D-3L)
Adverse events associated with post-operative analgesia | From surgey to discharge of hospital
  Catheter-related infection;Poor wound healing;Motor block;Drainage of operated joint

CONTACTS AND LOCATIONS:
Overall Officials: Min Su, MD., Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Losina E, Walensky RP, Kessler CL, Emrani PS, Reichmann WM, Wright EA, Holt HL, Solomon DH, Yelin E, Paltiel AD, Katz JN. Cost-effectiveness of total knee arthroplasty in the United States: patient risk and hospital volume. Arch Intern Med. 2009 Jun 22;169(12):1113-21; discussion 1121-2. doi: 10.1001/archinternmed.2009.136. PMID 19546411
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] Lieberman JR, Freiberg AA, Lavernia CJ. Practice management strategies among members of the American Association of Hip and Knee Surgeons. J Arthroplasty. 2012 Sep;27(8 Suppl):17-9.e1-6. doi: 10.1016/j.arth.2012.02.030. Epub 2012 Apr 12. PMID 22503334
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Wang H, Boctor B, Verner J. The effect of single-injection femoral nerve block on rehabilitation and length of hospital stay after total knee replacement. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):139-44. doi: 10.1053/rapm.2002.29253. PMID 11915059
- [Background] Paul JE, Arya A, Hurlburt L, Cheng J, Thabane L, Tidy A, Murthy Y. Femoral nerve block improves analgesia outcomes after total knee arthroplasty: a meta-analysis of randomized controlled trials. Anesthesiology. 2010 Nov;113(5):1144-62. doi: 10.1097/ALN.0b013e3181f4b18. PMID 20966667
- [Background] Carli F, Clemente A, Asenjo JF, Kim DJ, Mistraletti G, Gomarasca M, Morabito A, Tanzer M. Analgesia and functional outcome after total knee arthroplasty: periarticular infiltration vs continuous femoral nerve block. Br J Anaesth. 2010 Aug;105(2):185-95. doi: 10.1093/bja/aeq112. Epub 2010 Jun 14. PMID 20551021
- [Background] Ilfeld BM, Mariano ER, Girard PJ, Loland VJ, Meyer SR, Donovan JF, Pugh GA, Le LT, Sessler DI, Shuster JJ, Theriaque DW, Ball ST. A multicenter, randomized, triple-masked, placebo-controlled trial of the effect of ambulatory continuous femoral nerve blocks on discharge-readiness following total knee arthroplasty in patients on general orthopaedic wards. Pain. 2010 Sep;150(3):477-484. doi: 10.1016/j.pain.2010.05.028. Epub 2010 Jun 22. PMID 20573448
- [Background] Fischer HB, Simanski CJ, Sharp C, Bonnet F, Camu F, Neugebauer EA, Rawal N, Joshi GP, Schug SA, Kehlet H; PROSPECT Working Group. A procedure-specific systematic review and consensus recommendations for postoperative analgesia following total knee arthroplasty. Anaesthesia. 2008 Oct;63(10):1105-23. doi: 10.1111/j.1365-2044.2008.05565.x. Epub 2008 Jul 10. PMID 18627367
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Kazak Bengisun Z, Aysu Salviz E, Darcin K, Suer H, Ates Y. Intraarticular levobupivacaine or bupivacaine administration decreases pain scores and provides a better recovery after total knee arthroplasty. J Anesth. 2010 Oct;24(5):694-9. doi: 10.1007/s00540-010-0970-x. Epub 2010 Jun 23. PMID 20571832
- [Background] Koh IJ, Kang YG, Chang CB, Do SH, Seong SC, Kim TK. Does periarticular injection have additional pain relieving effects during contemporary multimodal pain control protocols for TKA?: A randomised, controlled study. Knee. 2012 Aug;19(4):253-9. doi: 10.1016/j.knee.2011.03.007. Epub 2011 Apr 19. PMID 21507661
- [Background] Lombardi AV Jr, Berend KR, Mallory TH, Dodds KL, Adams JB. Soft tissue and intra-articular injection of bupivacaine, epinephrine, and morphine has a beneficial effect after total knee arthroplasty. Clin Orthop Relat Res. 2004 Nov;(428):125-30. doi: 10.1097/01.blo.0000147701.24029.cc. PMID 15534532